CLINICAL TRIAL: NCT06344650
Title: Cellular, Molecular and Clinical Determinants of Bone Strength in in Vivo and Human Models of GH Excess. Cross-sectional and Prospective Study
Brief Title: Cellular, Molecular and Clinical Determinants of Bone Strength in in Vivo and Human Models of GH Excess.
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Fondazione Policlinico Universitario Campus Bio-Medico (Other); Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Andrea Giustina, Head of Endocrinology, IRCCS Ospedale San Raffaele
Other Study IDs: RF-2021-12373584
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood sample — Collection of blood serum for molecular and biochemical tests
Diagnostic Test: Radiological tests — Performance of radiological tests (DXA, VFA, TBS, BSi, HR-pQCT) and DXA morphometry
Other: Questionnaires — Compilation of questionnaires (AcroQol, SF-36)

SUMMARY:
Prospective observational clinical, molecular, translational study aimed at identifying the main determinants and predictive factors of fragility fracture risck in acromegaly patients

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of acromegaly
* availability to carry out outpatient checks
* ability to provide informed consent

Exclusion Criteria:

* Pregnancy
* use of glucocorticoids (except those in use for replacement therapy)
* alcohol abuse
* exacerbation of chronic disease
* serious comorbidities (renal or hepatic failure, heart attack, stroke)
* terminally ill, prolonged immobilization (>1 week)
* clinically evident fracture within the previous six months
* any other cause of secondary osteoporosis within the last five years
* any prolonged treatment with drugs with documented influence on bone metabolism during the previous 12 months, including treatment with antiresorptive or anabolic compounds for osteoporosis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acromegaly patients able to sign informed consent
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Identify the rate of morphometric vertebral fractures in acromegalic patients | 18 months
  Identify the rate of morphometric vertebral fractures in acromegalic patients 18 months after hospitalization for neurosurgery

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Giustina, Milan, Italy